CLINICAL TRIAL: NCT02319590
Title: The Role of Functional Active Anti-Angiotensin-Receptor 1 (ATR1)- and Anti-Endothelin-Receptor A (ETRA)-Antibodies and Autoreactive T Cells in Cardiomyopathy
Brief Title: Anti-Angiotensin-Receptor 1 (ATR1)-, Anti-Endothelin-Receptor A (ETRA)-Antibodies and T Cells in Cardiomyopathy
Acronym: T-CARD
Status: Completed | Type: Observational
Sponsor: Zurich Regional Health Center (Other)
Responsible Party: Principal Investigator, Urs Eriksson, Professor of Cardiology and Medicine, Chief Medical Office, Zurich Regional Health Center
Other Study IDs: 1
Record Dates: First submitted 2014-12-07; First posted 2014-12-18 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — T cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- heart failure, no CAD, QRS < 150ms: no CAD, QRS < 150ms
- heart failure, CAD QRS < 150ms: CAD, QRS < 150ms
- heart failure, CAD > 150ms: CAD, QRS > 150ms
- heart failure, no CAD, > 150ms: no CAD, QRS > 150ms

SUMMARY:
The study aims 1) to determine autoantibody titers against the AGTR1 receptor and against the ETA receptor, 2) to characterize cytokine expression profiles of heart-specific activated T cells in patients with systolic heart failure. Auto-antibody titers and specific cytokine expression profiles in heart-specific activated T cells will then be correlated with heart failure progression and outcome.

DETAILED DESCRIPTION:
1. AIM OF THE STUDY 1.1. Background Progressive interstitial fibrosis parallels pathological remodeling in the failing heart. This is particularly the case in patients with post-inflammatory dilated cardiomyopathy, but is also observed in ischemic and hypertensive heart disease. Both, Angiotensin II (AngII) and Endothelin-1 (ET1) induce the formation of the profibrotic cytokine TGFβ and promote fibrosis. From this point of view, it is not surprising that blocking the Renin-Angiotensin-Aldosterone-System (RAAS) evolved as key strategy to slow heart failure progression. Furthermore, recent data also points to an important role of Angiotensin II signaling in heart failure with preserved ejection fraction. In animal models, blocking the effect of AngII or ET1 reduces fibrotic remodeling following myocardial ischemia or in pulmonal hypertension. In line with these findings, we found no evidence of fibrotic remodeling in AGTR1-/- mice who recovered from acute myocarditis. Nevertheless, RAAS blockade is not efficient enough to completely prevent heart failure progression or even rapid deterioration in subgroups of the affected patients. Only recently, Riemekasten et al demonstrated that auto-antibodies against AGTR1 and ETAR are increased in systemic sclerosis and associated with increased pulmonary hypertension and lung fibrosis (2). Moreover, these auto-antibodies were shown to be functional active and to induce downstream expression of TGFβ -mRNA.

   Anti-AGTR1-Ab and Anti-ETAR-Ab might therefore directly promote fibrosis through activation of AGTR1 and ETAR. Furthermore, auto-reactive T-cells to the myosin heavy chain (MyHC) of the heart muscle were demonstrated to play an important role in both the initial inflammation during myocarditis as well as the progression of inflammation.

   1.2. Rationale for the current study Cardiac autoantibody titers are generally elevated in patients after myocardial infarction or suffering from systolic heart failure. In addition, we found experimental evidence for a critical role of AngII signaling in the development of cardiac fibrosis. We hypothesize that auto-immunological effects in general, and Anti-AGTR1-Ab, Anti- ETAR-Ab and auto-reactive T-cells in particular, are important and so far widely underestimated in the pathogenesis of cardiomyopathies and that they interfere with evidence based treatment approaches.

   1.3 Aims The objectives of this study are to
   * determine the concentration of Anti-AGTR1- and Anti-ETRA-AB in the patients blood.
   * determine the auto-reactive heart specific T-cells and their cytokine expression profile in patients blood.
   * to correlate these findings to outcome (hospitalizations due to heart failure, stroke, myocardial infarction, and death) and to cardiac function of the patient (VO2, Ejection fraction, NYHA class).
2. STUDY DESIGN Prospective pilot study.
3. PARTICITPANT ENTRY 3.1. Pre---registration evaluation Patients with cardiomyopathy and heart failure for 6 months or more will be recruited at the GZO Spital Wetzikon during ambulatory visits.
4. EFFICACY AND SAFETY VARIABLES 4.1. Efficacy variables and examinations 4.1.1 non---study specific variables and examinations Medical history

   * general information: age, gender, weight, height
   * actual medications
   * staging of heart failure according to the severty of symptoms and physical activity (New York Heart Association-classification) Electrocardiogram (ECG) For all electrocardiographic recordings a commercially available 12-lead ECG will be used and set at 25mm/s paper speed and 10mm/mV amplitude.

   Transthoracal echocardiography (TTE) TTE will be performed by a cardiologist. The following parameters will be recorded:
   * Left ventricular ejection fraction using Simpson Biplan method
   * Left ventricular end diastolic and end systolic diameter
   * Left atrial diameter
   * Peak velocity E, A; E/A quotient; TDI
   * Flow in pulmonary veines

   4.1.2 Study specific variables and examinations Determinations of Anti-AGTR1-AB and Anti-ETRA-AB Concentrations of Anti-AGTR1-AB and Anti-ETRA-AB will be measured using commercially available ELISA-Kits according to manufactures protocol (Celltrend, Luckenwalde, Germany).

   Evaluation of auto-reactive T-Cells Auto-reactive T-cells will be isolated from patient blood and analysed as described for organ-specificity (cMET+), for their reactivity against cardiac self-antigens and for their cytokine expression profile.
5. ASSESSMENT AND FOLLOW---UP The investigations during the visit are described in paragraph 4. The assessment are performed during the initial visit, at 4 months, and at 12 months.
6. STATISTICS AND DATA ANALYSIS As this is a pilot study and no published data on the observed parameters in cardiomyopathies are available, no power analysis was performed. Groups will be compared using ANOVA. Statistical significance will be assumed at a probability of p < 0.05.
7. REGULATORY ISSUES 7.1 Ethic approval The study will be conducted according to the current declaration of Helsinki, the Good Clinical Practice-guidelines and Swiss regulatory authority´s requirements. The study has been approved by the KEK (local ethics committee).

   7.2 Consent Written consent will be sought from participants only after full explanation of the study and time allowed for consideration. The right of the participant to refuse to participate without giving reasons will be respected. If the participant withdrawls his/her consent, data collected to the date of the withdrawal will be used.

   7.3 Confidentiality All study personnel will preserve the confidentiality of participants taking part in the study.

   7.4 Insurance Insurance is covered by "Zurich Versicherungsgesellschaft AG" for GZO Spital Wetzikon.
8. QUALITY CONTROL 8.1 Audits The investigators welcome audits by regulatory bodies to ensure adherence to GCP and regulatory requirements.

8.2 Data management A designated research nurse and/or research fellow will be responsible for data collection and data management.

8.3 Data privacy Access to personal data of participants is strictly limited to the investigators aforementioned. Raw data will be archieved for at least 10 years. Blood samples willbe analysed at the Center for Molecular Cardiology of the University of Zurich in the group for cardioimmunology and destroyed after definitive analysis. Blood sample collection will be done at GZO Spital Wetzikon. The blood samples will be anonymised directly after collection. All data sheets, blood samples and data fromanalysis will be anonymised to a two-digit code. The key to match the two-digit-code to the personal data of the patient will be stored in a separate, password-protected data base. Only the principal investigator and investigator Dr. med. Nazmi Krasniqi will have access to this data base.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 85
* Left ventricular ejection fraction <35%
* Established medical heart failure therapy
* Informed consent

Exclusion Criteria:

* mental or physical disability precluding informed consent or compliance with the protocol.
* Active auto-immune disease (rheumatoid arthritis, systemic sclerosis, sytemic lupus erythematodes, polymyositis or others)
* Active infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure patients, EF < 35%, either CAD (re-vascularized) or other type of heart failure
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-12; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of heart failure hospitalization, cardiovascular event, transplantation and death | 1 year
  cardiovascular event = cerebral ischemia/infarction, myocardial infarction/ACS, revascularization, critical limb/organ ischemia, vascular dissection, thromboembolism

SECONDARY OUTCOMES:
Ejection fraction (EF) | 1 Year
  Percentage end-diastolic blood volume ejected out of the left ventricle during systole; measured according to the modified Simpsons rule by echocardiography
Maximal Exercise Oxygen Consumption (VO2 max) | 6 month, 1 year
  Maximal Exercise Oxygen Consumption will be measured during treadmill exercise tests with simultaneous respiratory gas measurements (mL/min/kg).
NYHA class (NYHA) | 6 month, 1 year
  The New York Heart Association (NYHA) Functional Classification places patients in one of four categories based on how much they are limited during physical activity (NYHA class I, II, III, IV).
  I Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. no shortness of breath when walking, climbing stairs etc.
  II Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  III Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  IV Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Arrhythmia burden (AB) | 1 year
  Measured as numbers of relevant arrhythmias (ra), appropriate (as) and inappropriate shocks (ias) in ICD and CRT-D pts.
CRT Responder (CRT-Resp) | 1 year
  Measured as number of responding pts with CRT-D. Definition of responder: decrease in left ventricular end systolic volume of at least 30% (CRT-D pts only);

CONTACTS AND LOCATIONS:
Overall Officials: Urs Eriksson, MD, Principal Investigator — GZO Regional Health Center and University of Zurich
Locations (1):
- GZO Regional Health Center, Wetzikon, Switzerland